CLINICAL TRIAL: NCT04230148
Title: A Phase IV, Multi-center, Open-label Study to Determine the Safety, Tolerability and Clinical Outcomes Following Oral Administration of EGATEN™ (Triclabendazole) in Patients (6 Years of Age or Older) With Fascioliasis.
Brief Title: Study of Safety, Tolerability and Clinical Outcomes of Egaten in Fascioliasis Patients (6 Years of Age or Older).
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEGA230B2404
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Fascioliasis
Keywords: Acute Fascioliasis; Chronic Fascioliasis; Clinical Cure; Parasitological Cure; Egaten; Triclabendazole; Post-Marketing commitment
MeSH Terms: conditions — Fascioliasis | interventions — Triclabendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Egaten (Experimental): All subjects will receive Egaten as two 10 mg/kg doses given 12 hours apart.
  Interventions: Drug: Egaten (Triclabendazole) 250 mg tablets

INTERVENTIONS:
Drug: Egaten (Triclabendazole) 250 mg tablets — Egaten 250 mg scored tablets for oral use.
  Other Names: Triclabendazole

SUMMARY:
This is a multicenter, open label, non-comparative, single arm multi-country study in approximately 300 adult and pediatric subjects (≥ 6 years of age) with fascioliasis. The study population consists of male and female adult and pediatric patients (≥ 6 years of age). The study will enroll approximately 300 subjects with acute (minimum 15% of overall study population) or chronic fascioliasis. Enrolled subjects will receive two doses of 10 mg/kg of Egaten given approximately 12 hours apart. Subjects will be treated and followed up on an outpatient basis. After screening and post treatment, at Day 3 and Day 6 the subjects will be followed for safety and tolerability. These visits are primarily for safety follow up and may be telephonic or home visit by qualified personnel or onsite visits based on the investigator's discretion. During visits Day 10, Day 30, Day 60 and Day 90 post-treatment, the subjects will be followed for safety, tolerability and efficacy. On Day 15, Day 45 and Day 75, telephonic follow-up (primarily for safety) will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any study protocol specific assessment is performed.

   1. Parental/legal guardian informed consent must be obtained and signed for pediatric subjects (formally documented and witnessed, via an independent trusted witness) prior to any study related procedure.
   2. Subjects < 18 years old, who are capable of providing assent, must provide assent with parental/legal guardian consent or as per local ethical guidelines.
   3. If the subject is unable to read and write or otherwise incapable of signing an informed consent, then a witnessed consent according to local ethical standards is permitted.
2. Subjects (Adult and pediatric subjects ≥ 6 years of age and above 12.5 kg of weight) at time of consenting must have been diagnosed with fascioliasis based on clinical signs, symptoms and laboratory evaluations as per local clinical practice.

Exclusion Criteria:

1. Subjects diagnosed with ectopic fascioliasis, extrahepatic involvement (e.g., lungs, spleen, pancreas, subcutaneous tissue, gastrointestinal organs, etc.).
2. Subjects with known hypersensitivity to triclabendazole /other benzimidazole derivatives and/or any of the excipients in Egaten.
3. Subjects taking any anthelmintic medications within two weeks or 5 half-lives, whichever is longer prior to enrolling into study.
4. Inability or unwillingness to undergo study related procedures.
5. Subjects who in the judgment of the Clinical Investigator are unsuitable for the trial or who have to be excluded in order to be compliant with local fascioliasis management guidelines that may differ from the FDA approved label, including but not limited to :

   1. Subjects who are machine operators or drivers.
   2. Medical history of liver (other than fascioliasis), kidney or cardiac disease.
6. Females (including under the age of 18) known to be pregnant or testing positive for pregnancy at screening.
7. Lactating women unwilling to discontinue lactation up to 72 hours after the second dose administration or as per local guidelines.
8. Subjects requiring therapeutic drug monitoring of CYP2C19 substrate(s) (e.g. S-mephenytoin).
9. Subjects with medical history of QT prolongation or a history of symptoms compatible with a long QT interval or on medication which prolong the QT interval.

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2026-03-29 (Estimated); Study Completion 2026-03-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with On-Treatments Adverse Events, Serious Adverse Events, and Deaths | Day 90
  Analysis of absolute and relative frequencies for treatment emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths by primary System Organ Class (SOC) to demonstrate that Egaten administered as two 10 mg/kg doses given 12 hours apart in subjects with Fascioliasis is safe through the monitoring of relevant clinical and laboratory safety parameters.

SECONDARY OUTCOMES:
Clinical cure rate in Acute Fascioliasis subjects over time. | Day 10, Day 30, Day 60 and Day 90
  The clinical cure rate in Acute Fasciolisis subjects will be measured by the proportion of subjects with:
  1. Resolution of baseline signs and symptoms.
  2. Improvement in baseline laboratory parameters.
  3. Improvement in baseline ultrasound findings.
Parasitological cure rate in Chronic Fascioliasis subjects over time. | Day 10, Day 30, Day 60 and Day 90
  The parasitological cure rate in Chronic Fascioliasis subjects will be measured by the proportion of subjects with absence of fasciola eggs confirmed by stool examination.
Clinical cure rate of Chronic Fascioliasis subjects over time. | Day 10, Day 30, Day 60 and Day 90
  The clinical cure rate in Chronic Fasciolisis subjects will be measured by the proportion of subjects with:
  1. Resolution of baseline signs and symptoms.
  2. Improvement in baseline laboratory parameters.
  3. Improvement in baseline ultrasound findings.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Novartis Investigative Site, Medellín, Antioquia, Colombia
- Egypt (2):
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
- Peru (2):
  - Novartis Investigative Site, San Martín de Porres, Lima region
  - Novartis Investigative Site, Cusco
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Gaziantep, Sehitkamil
  - Novartis Investigative Site, Sur
  - Novartis Investigative Site, Van
- Novartis Investigative Site, Qui Nhon, Binh Dinh, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com